CLINICAL TRIAL: NCT01272050
Title: Dose Intensified Salvage Radiotherapy in Biochemically Relapsed Prostate Cancer Without Macroscopic Disease. A Randomized Phase III Trial.
Brief Title: Radiation Therapy in Treating Patients With Relapsed Prostate Cancer After Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Swiss Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: SAKK 09/10; SWS-SAKK-09/10; EU-21088; CDR0000691926 (Other: NCI)
Record Dates: First submitted 2011-01-06; First posted 2011-01-07 (Estimated); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Prostate Cancer
Keywords: adenocarcinoma of the prostate; recurrent prostate cancer; stage IIA prostate cancer; stage IIB prostate cancer; stage III prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A: 64 Gy - Radiation Therapy (Active Comparator): Arm A: 64 Gy (32 x 2 Gy) without hormonal treatment
  Interventions: Radiation: radiation therapy
- Arm B: 70 Gy - Radiation Therapy (Active Comparator): Arm B: 70 Gy (35 x 2 Gy) without hormonal treatment
  Interventions: Radiation: radiation therapy

INTERVENTIONS:
Radiation: radiation therapy — RT in the standard arm A will be administered to a total dose of 64 Gy in 32 fractions of 2 Gy over 6.4 weeks. RT in the experimental arm B will be administered to a total dose of 70 Gy in 35 fractions of 2 Gy over 7 weeks.
  Megavoltage equipments with nominal photon energies ≥ 6 MV are required. Rotational techniques such as Tomotherapy®, Rapidarc®, intensity-modulated arc technique (IMAT) and volumetric-modulated arc therapy (VMAT) will also be eligible. The patient will be treated in an isocentric setting and all fields will be applied for 5 days per week for the total RT duration.

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to kill tumor cells. It is not yet known which radiation therapy regimen is more effective in treating patients with relapsed prostate cancer.

PURPOSE: This randomized phase III trial is studying the side effects of radiation therapy and comparing two radiation therapy regimens in treating patients with relapsed prostate cancer after surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

* To determine the tumor control in patients with biochemically relapsed prostate cancer without macroscopic disease treated with dose-intensive salvage radiotherapy.
* To determine the toxicity in these patients.
* To determine the quality of life of these patients.

OUTLINE: This is a multicenter study. Patients are stratified according to Gleason score (≥ 8 vs 7 vs ≤ 6), pathological tumor classification (pT3b vs others), lymphadenectomy performed (yes [pN0] vs no [cN0]), persistent PSA after prostatectomy (detectable [≥ 0.1 ng/mL] vs undetectable [< 0.1 ng/mL]), PSA at randomization (> 0.5 ng/mL vs ≤ 0.5 ng/mL), participating center, and radiotherapy technique (3-dimensional conformal radiation therapy [3D-CRT] vs intensity-modulated radiation therapy [IMRT]/rotational techniques). Patient are randomized to 1 of 2 treatment arms.

* Arm A: Beginning at least 12 weeks after surgery, patients undergo radiotherapy* once a day, 5 days a week, for 6.4 weeks for a total dose of 64 Gy (in 32 fractions of 2 Gy over 6.4 weeks).
* Arm B: Patients undergo radiotherapy* once a day, 5 days a week, for 7 weeks for a total dose of 70 Gy (in 35 fractions of 2 Gy over 7 weeks).

NOTE: *3-dimensional conformal radiation therapy, rotational techniques such as Tomotherapy®, Rapidarc®, or intensity-modulated arc technique and volumetric-modulated arc therapy are all eligible.

Patients complete quality-of-life questionnaires at baseline and at 3, 12, 24, 36, 48, and 60 months after completing study therapy.

After completion of study treatment, patients are followed every 6 months for 3 years and then every 12 months for up to 10 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of adenocarcinoma of the prostate

  * Lymph node negative disease

    * Stage pT2a-3b; R0-1; pN0 or cN0
* Undergone a radical prostatectomy ≥ 12 weeks prior to randomization
* PSA progression after prostatectomy defined as two consecutive rises with the second rising value > 0.1 ng/mL OR three consecutive rises (the first value must be measured 4 weeks after radical prostatectomy)
* PSA ≤ 2 ng/mL at randomization

  * No persistent PSA > 0.4 ng/mL, 4-20 weeks after radical prostatectomy
* No palpable prostatic fossa mass suggestive of recurrence, unless an ultrasound-guided biopsy is non-malignant
* No pre-salvage radiotherapy pelvic lymph node enlargement > 1 cm in short axis diameter of the abdomen and pelvis (cN1) (unless the enlarged lymph node is sampled and negative)
* No evidence of macroscopic local recurrence or metastatic disease on pre-salvage radiotherapy MRI (with IV contrast) or multislice computed tomography (with IV and oral contrast) of the abdomen and pelvis assessed within 16 weeks prior to randomization
* No presence or history of bone metastases (bone scan must be performed in case of clinical suspicion [e.g., bone pain])
* Gleason score must be available

PATIENT CHARACTERISTICS:

* WHO performance status 0-1
* Fertile patients must use effective contraception during and for 6 months after completion of study therapy
* Compliant and geographically proximal to allow for proper staging and follow-up
* No prior invasive malignancy, except non-melanomatous skin cancer or other malignancies with a documented disease-free survival of ≥ 5 years
* No bilateral hip prosthesis
* No severe or active co-morbidity likely to impact on the advisability of dose-intensive salvage radiotherapy, including any of the following:

  * History of inflammatory bowel disease
  * Acute bacterial or fungal infection requiring intravenous antibiotics at the time of randomization
  * Unstable angina and/or congestive heart failure requiring hospitalization within the past 6 months
  * Transmural myocardial infarction within the past 6 months
  * Chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy at the time of randomization
* No psychiatric disorder precluding understanding of information on trial-related topics, giving informed consent, or filling out quality-of-life questionnaires

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No prior pelvic radiotherapy
* No hormonal treatment or bilateral orchiectomy prior to or following prostatectomy
* At least 4 weeks since prior and no concurrent use of products known to affect PSA levels (e.g., PC Calm, PC Plus, PC SPES, finasteride, or fluconazole)
* At least 30 days since prior treatment in another clinical trial
* No other concurrent anticancer treatments, including luteinizing hormone-releasing hormone (LHRH) analogues, antiandrogens, orchiectomy, or chemotherapy
* No other concurrent investigational or experimental treatments or drugs

INCLUSION CRITERIA

* Patient must give written informed consent before randomization.
* Lymph node negative adenocarcinoma of the prostate treated with radical prostatectomy at least 12 weeks before randomization. Tumor stage pT2a-3b, R0-1, pN0 or cN0 according to the UICC TNM 2009 (see Appendix 1), Gleason score available.
* PSA progression after prostatectomy defined as two consecutive rises with the final PSA > 0.1 ng/mL or three consecutive rises. The first value must be measured earliest 4 weeks after radical prostatectomy.
* PSA at randomization ≤ 2 ng/mL.
* WHO performance status 0-1 at randomization.
* Age at randomization between 18 and 75 years.
* Baseline QoL questionnaire (QLQ) has been completed.
* Patient agrees not to father a child during salvage RT and during 6 months thereafter.
* Patient compliance and geographic proximity allow proper staging and follow-up.
* The responsible pathologist has agreed to provide sample material for central pathological review (see Section 16) and tissue banking (only if patient gave informed consent) within the specified timelines.

EXCLUSION CRITERIA

* Persistent PSA 4-20 weeks after radical prostatectomy > 0.4 ng/mL
* Palpable prostatic fossa mass suggestive of recurrence, unless an ultrasound guided biopsy is non-malignant.
* Pre-salvage RT pelvic lymph node enlargement > 1 cm in short axis diameter of the abdomen and pelvis (cN1), unless the enlarged lymph node is sampled and negative, and/or evidence of macroscopic local recurrence or metastatic disease on pre-salvage RT MRI (magnetic resonance imaging; with i.v. contrast) or multislice computed tomography (CT; with i.v. and oral contrast) of the abdomen and pelvis assessed within 16 weeks prior to randomization.
* Presence or history of bone metastases. Bone scan must be performed in case of clinical suspicion (e.g. bone pain).
* Prior invasive malignancy, except non-melanomatous skin cancer or other malignancies with a documented disease-free survival for a minimum of 5 years.
* Hormonal treatment or bilateral orchiectomy prior to or following prostatectomy.
* Bilateral hip prosthesis.
* Prior pelvic radiotherapy.
* The use of products known to affect PSA levels within 4 weeks prior to start of trial treatment (e.g. PC Calm, PC Plus, PC SPES, finasteride, fluconazole).
* Severe or active co-morbidity likely to impact on the advisability of dose intensified salvage RT.
* Psychiatric disorder precluding understanding of information on trial related topics, giving informed consent or filling out QoL questionnaires.
* Concurrent treatment with other experimental drugs or other anti-cancer therapy, treatment in a clinical trial within 30 days prior to trial entry.

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Actual)
Dates: Start 2011-01-06 (Actual); Primary Completion 2020-07-03 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
Freedom from biochemical progression | from the day of trial randomization to the day of either first recorded biochemical progression, clinical progression or death due to clinical progression up to 10 years.

SECONDARY OUTCOMES:
Clinical progression-free survival | from the day of randomization to the day of the first record of either local or regional recurrence, distant recurrence, start of hormonal treatment, or death due to any cause up to 10 years.
Time to hormonal treatment | time from trial randomization to start of hormonal treatment up to 10 years.
Prostate cancer-specific survival | time from trial randomization to the date of death due to prostate cancer up to 10 years.
Overall survival | time from trial randomization to the date of death from any cause up to 10 years.
Acute and late gastrointestinal and genitourinary toxicity according to CTCAE v 4.0 | occurring during treatment and up to 3 months after completion of treatment. Late toxicity is defined as occurring later than 3 months after end of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Pirus Ghadjar, MD, Study Chair — Charite University, Berlin, Germany; Daniel M. Aebersold, Prof., Study Chair — Bern University Hospital; George N. Thalmann, Prof., Study Chair — Bern University Hospital; Daniel Zwahlen, PD Dr., Study Chair — Kantonsspital Graubünden
Locations (28):
- Belgium (3):
  - Ziekenhuis Netwerk Antwerpen Middelheim, Antwerp
  - Ghent University Hospital, Ghent
  - St. Lukas Hospital Ghent, Ghent
- Germany (11):
  - Universitaetsklinikum Aachen, Klinik für Strahlentherapie, Aachen
  - Charite University Hospital - Campus Virchow Klinikum, Berlin
  - University Hospital and Medical Faculty Technical University of Dresden, Dresden
  - Universitaetsklinikum Essen, Klinik für Strahlentherapie, Essen
  - Universitätsklinikum Saarland, Homburg
  - Klinikum der LMU Muenchen, Munich
  - Technische Universitaet Muenchen, Munich
  - Klinikum der Universitaet Regensburg, Regensburg
  - Klinik und Poliklinik fuer Strahlentherapie - Universitaetsklinikum Rostock, Rostock
  - Universitaet Tuebingen, Tübingen
  - Klinik fuer Strahlentherapie Universitaet Wuerzburg, Würzburg
- Switzerland (14):
  - Kantonsspital Aarau, Aarau
  - Universitaetsspital-Basel, Basel
  - Istituto Oncologico della Svizzera Italiana - Ospedale Regionale Bellinzona e Valli, Bellinzona
  - Inselspital Bern, Bern
  - Radio-Onkologiezentrum Biel-Seeland-Berner Jura AG, Biel
  - Kantonsspital Graubuenden, Chur
  - Kantonsspital Luzern, Lucerne
  - Kantonsspital Muensterlingen, Münsterlingen
  - Kantonsspital - St. Gallen, Sankt Gallen
  - Hopital de Sion, Sion
  - Radio-Onkologie Berner Oberland AG, Thun
  - Klinik Hirslanden, Zurich
  - City Hospital Triemli, Zurich
  - UniversitaetsSpital Zuerich, Zurich

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ghadjar P, Hayoz S, Zwahlen DR, Holscher T, Arnold W, Polat B, Hildebrandt G, Hoffmann E, Plasswilm L, Papachristofilou A, Schar C, Sumila M, Zaugg K, Guckenberger M, Ost P, Reuter C, Bosetti DG, Khanfir K, Riesterer O, Beck M, Thalmann GN, Aebersold DM; Swiss Group for Clinical Cancer Research (SAKK). Dose-intensified Versus Conventional-dose Salvage Radiotherapy for Biochemically Recurrent Prostate Cancer After Prostatectomy: Long-term Data from the SAKK 09/10 Randomised Phase 3 Trial. Eur Urol. 2026 Jan 5:S0302-2838(25)04875-4. doi: 10.1016/j.eururo.2025.12.020. Online ahead of print. PMID 41494929
- [Derived] Zwahlen DR, Schroder C, Holer L, Bernhard J, Holscher T, Arnold W, Polat B, Hildebrandt G, Muller AC, Martin Putora P, Papachristofilou A, Schar C, Hayoz S, Sumila M, Zaugg K, Guckenberger M, Ost P, Giovanni Bosetti D, Reuter C, Gomez S, Khanfir K, Beck M, Thalmann GN, Aebersold DM, Ghadjar P. Erectile function preservation after salvage radiation therapy for biochemically recurrent prostate cancer after prostatectomy: Five-year results of the SAKK 09/10 randomized phase 3 trial. Clin Transl Radiat Oncol. 2024 Apr 25;47:100786. doi: 10.1016/j.ctro.2024.100786. eCollection 2024 Jul. PMID 38706726
- [Derived] Beck M, Sassowsky M, Schar S, Mathier E, Halter M, Zwahlen DR, Holscher T, Arnold W, Polat B, Hildebrandt G, Muller AC, Putora PM, Papachristofilou A, Hayoz S, Schar C, Li Q, Sumila M, Zaugg K, Guckenberger M, Ost P, Bosetti DG, Reuter C, Gomez S, Khanfir K, Aebersold DM, Ghadjar P, Pra AD. Adherence to Contouring and Treatment Planning Requirements Within a Multicentric Trial: Results of the Quality Assurance of the SAKK 09/10 trial. Int J Radiat Oncol Biol Phys. 2022 May 1;113(1):80-91. doi: 10.1016/j.ijrobp.2021.12.174. Epub 2022 Jan 3. PMID 34990777
- [Derived] Ghadjar P, Hayoz S, Bernhard J, Zwahlen DR, Holscher T, Gut P, Polat B, Hildebrandt G, Muller AC, Plasswilm L, Papachristofilou A, Schar C, Sumila M, Zaugg K, Guckenberger M, Ost P, Reuter C, Bosetti DG, Khanfir K, Gomez S, Wust P, Thalmann GN, Aebersold DM; Swiss Group for Clinical Cancer Research (SAKK). Dose-intensified Versus Conventional-dose Salvage Radiotherapy for Biochemically Recurrent Prostate Cancer After Prostatectomy: The SAKK 09/10 Randomized Phase 3 Trial. Eur Urol. 2021 Sep;80(3):306-315. doi: 10.1016/j.eururo.2021.05.033. Epub 2021 Jun 14. PMID 34140144
- [Derived] Ghadjar P, Hayoz S, Bernhard J, Zwahlen DR, Holscher T, Gut P, Guckenberger M, Hildebrandt G, Muller AC, Plasswilm L, Papachristofilou A, Stalder L, Biaggi-Rudolf C, Sumila M, Kranzbuhler H, Najafi Y, Ost P, Azinwi NC, Reuter C, Bodis S, Kaouthar K, Wust P, Thalmann GN, Aebersold DM. Acute Toxicity and Quality of Life After Dose-Intensified Salvage Radiation Therapy for Biochemically Recurrent Prostate Cancer After Prostatectomy: First Results of the Randomized Trial SAKK 09/10. J Clin Oncol. 2015 Dec 10;33(35):4158-66. doi: 10.1200/JCO.2015.63.3529. Epub 2015 Nov 2. PMID 26527774